CLINICAL TRIAL: NCT00319995
Title: Efficacy and Safety of Combination Loratadine/Montelukast QD vs Pseudoephedrine and Placebo in the Treatment of Subjects With Seasonal Allergic Rhinitis
Brief Title: Effects of Loratadine/Montelukast vs Pseudoephedrine and Placebo in Patients With Seasonal Allergic Rhinitis (Study P04095) (COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04095; Doc ID 3058224;; SCH 445761
Record Dates: First submitted 2006-04-28; First posted 2006-04-27 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Loratadine; montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: loratadine; montelukast

SUMMARY:
This is a Phase 3, randomized, parallel-group, multicenter, double-dummy, double-blind study with a screening period. Subjects will receive one of the following three treatment groups for 15 days: loratadine 10 mg/montelukast 10 mg combination, pseudoephedrine 240 mg, or placebo. The primary objective of this study is to assess the efficacy of the combination of loratadine/montelukast, a once-daily tablet containing 10 mg loratadine and 10 mg montelukast, compared with placebo in subjects with seasonal allergic rhinitis (SAR) in relieving the symptom of nasal congestion. The safety profile of combined loratadine/montelukast relative to placebo and pseudoephedrine will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 years or older, of either sex and of any race.
* At least a 2-year documented history of SAR with symptoms during the study season.
* A positive skin-prick test response to seasonal
* Clinically symptomatic at Screening and at the Baseline Visits
* General good health.
* Freedom from any clinically significant disease, other than SAR, that would interfere with the study evaluations.
* Willingness (subjects and/or a parent/guardian) to give written informed consent and ability to adhere to dosing and visit schedules and meet study requirements.
* Negative pregnancy test

Exclusion Criteria:

* A history of anaphylaxis and/or other severe local reaction(s) to skin testing.
* Asthma requiring chronic use of inhaled or systemic corticosteroids.
* Current or history of frequent, clinically significant sinusitis or chronic purulent postnasal drip.
* Rhinitis medicamentosa.
* A history of allergies to more than two classes of medications or allergy to or intolerance of antihistamines, montelukast, or pseudoephedrine.
* An upper respiratory tract or sinus infection that required antibiotic therapy without at least a 14 day washout prior to the Screening Visit, or a viral upper respiratory infection within 7 days before the Screening Visit.
* Nasal structural abnormalities, including large nasal polyps and marked septal deviations, that significantly interfere with nasal air flow.
* Dependence (in the opinion of the investigator) on nasal, oral, or ocular decongestants, nasal topical antihistamines, or nasal steroids.
* Narrow-angle glaucoma, increased intraocular pressure, urinary retention, hypertension, severe coronary artery disease, ischemic heart disease, diabetes mellitus, hyperthyroidism, renal impairment, or prostatic hypertrophy, and those receiving monamine oxidase (MAO) inhibitor therapy.
* Use of any drug in an investigational protocol in the 30 days before the Screening Visit.
* Current immunotherapy (desensitization therapy), unless on a regular maintenance schedule prior to the Screening Visit, which should be maintained for the remainder of the study. No desensitization treatment within 24 hours before any visit.
* Requirement for chronic use of tricyclic antidepressants.
* Pregnancy or lactation.
* Family member of the investigation study staff.
* Current evidence of clinically significant hematopoietic, cardiovascular, hepatic, renal, neurologic, psychiatric, autoimmune disease, or other disease that precludes the subject's participation in the study. Particular attention should be given to exclude subjects with conditions that would currently interfere with the absorption, distribution, metabolism, or excretion of the study drug or interfere with the subject's ability to complete or reliably complete the diary card.
* Significant medical condition(s) that, in the judgment of the investigator, might interfere with the study or require treatment.
* Compromised ability to provide informed consent..
* A history of noncompliance with medications or treatment protocols.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1095 (Actual)
Dates: Start 2006-03-01 (Actual); Primary Completion 2006-06-01 (Actual); Study Completion 2006-06-28 (Actual)

REFERENCES:
- [Derived] Prenner B, Anolik R, Danzig M, Yao R. Efficacy and safety of fixed-dose loratadine/montelukast in seasonal allergic rhinitis: effects on nasal congestion. Allergy Asthma Proc. 2009 May-Jun;30(3):263-9. doi: 10.2500/aap.2009.30.3228. PMID 19549427